CLINICAL TRIAL: NCT00968617
Title: A Phase IIb Randomized, Active Comparator-Controlled, Open-Label Clinical Trial to Study the Efficacy and Safety of MK2578 for the Treatment of Anemia in ESA (Erythropoiesis-Stimulating Agent)-Naive Patients With Chronic Kidney Disease Who Are Not on Dialysis.
Brief Title: A Study of MK2578 in Patients With Chronic Kidney Disease Who Are Not on Dialysis (2578-002)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2578-002; 2009_653
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: Anemia
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK2578 1.0 mcg/kg (Experimental): MK2578
  Interventions: Drug: MK2578
- MK2578 2.0 mcg/kg (Experimental): MK2578
  Interventions: Drug: MK2578
- MK2578 3.6 mcg/kg (Experimental): MK2578
  Interventions: Drug: MK2578
- Darbepoetin alfa (Active Comparator): darbepoetin alfa
  Interventions: Drug: Comparator: darbepoetin alfa

INTERVENTIONS:
Drug: MK2578 — MK2578 1.0 mcg/kg/month
  Arms: MK2578 1.0 mcg/kg
Drug: MK2578 — MK2578 2.0 mcg/kg/month
  Arms: MK2578 2.0 mcg/kg
Drug: MK2578 — MK2578 3.6 mcg/kg/month
  Arms: MK2578 3.6 mcg/kg
Drug: Comparator: darbepoetin alfa — darbepoetin alfa
  Arms: Darbepoetin alfa

SUMMARY:
This study will define an effective starting dose for subcutaneous administration of MK2578 to correct anemia in erythropoiesis-stimulating agent (ESA)-naive patients with chronic kidney disease (CKD) who are not on dialysis while evaluating its safety.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or is a female who either cannot have children or who agrees to use appropriate contraceptive measures
* Patient has chronic kidney disease

Exclusion Criteria:

* Patient is morbidly obese
* Patient has used another erythropoiesis (red blood cell formation) stimulating agent within 12 weeks of screening
* Patient will require dialysis during the study or is planning to have a kidney transplant within the next 6 months
* Patient has had a blood transfusion within 12 weeks of screening
* Patient has had major surgery within the past 12 weeks or plans to have surgery
* Patient has Human Immunodeficiency Virus (HIV)
* Patient has a history of diseases other than CKD known to cause anemia
* Patient has severe congestive heart failure
* Patient has history of malignant cancer, except certain skin or cervical cancers
* Patient has a history of grand mal seizures within the last 6 months
* Patient is pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in Cohorts 1 and 2 were to receive 1.0 mcg/kg/month and 2.0 mcg/kg/month, respectively, of MK2578. Participants in Cohort 3 were to be randomized to MK2578 3.6 mcg/kg/month or to weekly doses of darbepoetin alfa 0.45 mcg/kg/week. Cohort 1 was the only cohort initiated.
Groups:
- MK2578: MK2578 1.0 mcg/kg given subcutaneously (SC) every month.
Period: Overall Study
Arm/Group | MK2578
Started | 7
Completed | 1
Not Completed | 6
Not completed — Study terminated by sponsor | 6

BASELINE CHARACTERISTICS:
Arm/Group | MK2578
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin Level at Week 4
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | MK2578
Number analyzed (Participants) | 7
g/dL
  Baseline Hemoglobin | 9.3 (0.4)
  Change from Baseline in Hemoglobin at Week 4 | 0.5 (0.4)

2. Primary Outcome: Number of Participants With Composite Events of Death, Myocardial Infarction and Cerebrovascular Accident, Serious Events of Unstable Angina, Transient Ischemic Attack, Arrythmia and Congestive Heart Failure, Peripheral Thrombo-embolic Events
Time Frame: 16 Weeks
Measure: Number; unit: Participants
Arm/Group | MK2578
Number analyzed (Participants) | 7
Participants | 0

3. Primary Outcome: Number of Participants With Composite Events of Transfusion-related Adverse Experiences
Time Frame: 16 Weeks
Measure: Number; unit: Participants
Arm/Group | MK2578
Number analyzed (Participants) | 7
Participants | 0

4. Primary Outcome: Number of of Participants With Composite Events of Injection Site Reactions
Time Frame: 16 Weeks
Measure: Number; unit: Participants
Arm/Group | MK2578
Number analyzed (Participants) | 7
Participants | 1

5. Primary Outcome: Number of Participants With Hypertension, Seizure, and Pure Red Cell Aplasia
Time Frame: 16 Weeks
Measure: Number; unit: Participants
Arm/Group | MK2578
Number analyzed (Participants) | 7
Participants
  Hypertension | 1
  Seizure | 0
  Pure red cell aplasia | 0

6. Primary Outcome: Number of Participants With Confirmed, Treatment Emergent Antibodies to MK2578
Time Frame: 16 Weeks
Measure: Number; unit: Participants
Arm/Group | MK2578
Number analyzed (Participants) | 7
Participants | NA — Immunogenicity assays for antibodies to MK2578 were not performed due to early study termination.

7. Secondary Outcome: Hemoglobin Concentration After Treatment With MK2578
Time Frame: Weeks 1-10 and Week 12
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | MK2578
Number analyzed (Participants) | 7
g/dL
  Week 1 (n=6) | 9.2 (0.8)
  Week 2 (n=5) | 9.8 (0.6)
  Week 3 (n=5) | 9.9 (0.7)
  Week 4 (n=7) | 9.8 (0.6)
  Week 5 (n=5) | 10.3 (0.7)
  Week 6 (n=4) | 10.4 (0.8)
  Week 7 (n=3) | 10.8 (0.9)
  Week 8 (n=4) | 11.1 (0.7)
  Week 9 (n=2) | 10.9 (0.4)
  Week 10 (n=1) | 10.6 (NA) — No standard deviation exists for n=1.
  Week 12 (n=1) | 11.1 (NA) — No standard deviation exists for n=1.

8. Secondary Outcome: Change From Baseline in Hemoglobin Level
Time Frame: Weeks 1-3, 5-10, and Week 12
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | MK2578
Number analyzed (Participants) | 7
g/dL
  Change from Baseline in Hemoglobin at Week 1 (n=6) | -0.1 (0.6)
  Change from Baseline in Hemoglobin at Week 2 (n=5) | 0.5 (0.4)
  Change from Baseline in Hemoglobin at Week 3 (n=5) | 0.6 (0.7)
  Change from Baseline in Hemoglobin at Week 5 (n=5) | 0.9 (0.4)
  Change from Baseline in Hemoglobin at Week 6 (n=4) | 1.0 (0.6)
  Change from Baseline in Hemoglobin at Week 7 (n=3) | 1.3 (0.7)
  Change from Baseline in Hemoglobin at Week 8 (n=4) | 1.6 (0.4)
  Change from Baseline in Hemoglobin at Week 9 (n=2) | 1.5 (0.1)
  Change from Baseline in Hemoglobin at Week 10(n=1) | 1.6 (NA) — No standard deviation exists for n=1.
  Change from Baseline in Hemoglobin at Week 12(n=1) | 2.1 (NA) — No standard deviation exists for n=1.

9. Secondary Outcome: Number of Participants Who Were Responders
Description: Responder was defined as a participant achieving (pre-transfusion) an increase from baseline hemoglobin of greater than or equal to 1 g/dL and a hemoglobin concentration of greater than or equal to 11 g/dL.
Time Frame: Each week up to 12 weeks
Measure: Number; unit: Participants
Arm/Group | MK2578
Number analyzed (Participants) | 7
Participants | 4

ADVERSE EVENTS:
Arm/Group | MK-2578
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2578 (N=7)
Tachycardia (Cardiac disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Cohort 1 (MK2578 1.0 mcg/kg) was the only cohort initiated because the study was prematurely terminated by the sponsor. 7 participants received at least 1 dose of MK2578 & 2 participants received all 3 doses. Data presented are for Cohort 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.